CLINICAL TRIAL: NCT03699111
Title: Identification of New Patient Stratification Tools in Microsatellite Stable (MSS) RAS mt Metastatic Colorectal Cancer (mCRC) - COLOSSUS
Brief Title: Identification of New Patient Stratification Tools in MSS RAS mt mCRC
Acronym: COLOSSUS
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: CTRIAL-IE 17-26
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a translational, multicentre and multinational study. The aim of this study is to identify new patient stratification tools in microsatellite stable RAS mutant metastatic Colorectal Cancer

DETAILED DESCRIPTION:
The rational of COLOSSUS is to provide new and more effective stratification tools and therapeutic interventions, specifically tailored to MSS RAS mt mCRC patients

ELIGIBILITY:
Inclusion criteria

Patient Status

1. Ability to give signed informed consent prior to any study specific procedures and willing and able to comply with the protocol,
2. Age ≥ 18 years,
3. ECOG status of ≤ 2,
4. At least 16 weeks of life expectancy at time of entry into the study.

   Disease-related
5. Histologically confirmed stage IV MSS RAS mt mCRC as per standard diagnostic tests,
6. Unresectable and measurable disease (at least one measurable target lesion) as per clinical and radiologic criteria (RECIST v.1.1),
7. No prior chemotherapy and/or radiation therapy for CRC administered in the metastatic setting,
8. Scheduled to receive or receiving SOC chemotherapy with fluoropyrimidines and oxaliplatin +/- bevacizumab (baseline blood sample should be collected and questionnaires completed during pre-screening and before chemotherapy initiation),
9. Availability of archival formalin-fixed paraffin-embedded (FFPE) tissue from:

   1. Preferred: surgical resection of the primary or metastatic tumour

      or
   2. Biopsy samples (biopsy taken at endoscope, needle core or surgical incision or excision) obtained from the primary or metastatic tumour.

The archival FFPE tissue blocks must be obtained during initial diagnosis (before patient was exposed to any chemotherapy and/or radiation therapy).

Exclusion Criteria

1. Patient with CRC that has received any therapy for CRC before:

   1. surgical resection of tissue that would be utilised in this study

      or
   2. biopsy procedure for tissue that would be utilised in this study,
2. Patient who has received any investigational product within 28 days of the first day of palliative chemotherapy administration,
3. Patient with any significant history of non-compliance to medical treatments or with inability to grant reliable informed consent,
4. Patient with clinical or laboratory contraindication to receive SOC chemotherapy with fluoropyrimidines and oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with stage IV MSS RAS mutant colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Stratification Tools | 4 years
  Identification and technical (analytical) validation of new patient stratification tools (COLOSSUS subtypes) in MSS RAS mt mCRC using a novel integrative systems biomedicine multi-omics discovery framework.

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (3):
  - Private Practice Oncology, Heidelberg, Heidelberg
  - University Hospital, Mannheim, Mannheim
  - Private Practice Oncology, Speyer, Speyer
- Ireland (5):
  - Bon Secours Hospital, Cork, Cork
  - Beaumont Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided